CLINICAL TRIAL: NCT00867399
Title: A Multiple Dose Study of Safety, Tolerability and Pharmacokinetics of ABT-126 in Elderly Subjects
Brief Title: A Safety and Tolerability Study of ABT-126 in Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Llano, MD, PhD, Associate Medical Director, Abbott
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M10-717
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 20mg of ABT-126 QD (Active Comparator): 20 mg of ABT-126 QD for 10 days
  Interventions: Drug: ABT-126
- 30mg and 45mg ABT-126 QD (Active Comparator): 30 mg and 45mg of ABT-126 QD for 21 days
  Interventions: Drug: ABT-126

INTERVENTIONS:
Drug: ABT-126 — See arm for details

SUMMARY:
The objectives of this study are to assess the safety, tolerability and pharmacokinetics of ABT-126 in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 65 years or greater.
* Has a MMSE score of 27 or higher.

Exclusion Criteria:

* History of dementia including by not limited to Alzheimer's disease, Parkinson's disease and mult-infarct dementia.
* History of any significant neurological disease.
* Has an estimated creatinine clearance < 30 mL/min

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessments (i.e., ECG, clinical laboratory tests, vital signs, weight, AE assessment, physical and brief neurological examinations) | Study Days -1 thru Day 28
Assess the Pharmacokinetics | Study Days -1 thru Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 17283, Orlando, Florida, United States